CLINICAL TRIAL: NCT04487730
Title: Social Reward and Its Effect on Brain Functions in Psychotherapies for Mid- and Late-Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-04021860; K23MH123864-01 (NIH)
Record Dates: First submitted 2020-07-23; First posted 2020-07-27 (Actual); Results first posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Late Life Depression; Psychotherapy; Mechanisms of Action; Positive Valence System; Social Reward
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial. Participants will be randomly assigned to 9-weeks of either "Engage-S" Psychotherapy or "Symptom Review and Psychoeducation" (SRP) Psychotherapy
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Engage & Connect" Psychotherapy (Experimental): "Engage & Connect", a modified adapted version of "Engage". Its principal intervention is "social reward exposure" - facilitating engagement in rewarding and meaningful social activities with significant others. In "Engage-S" therapy, individuals with depression work with a therapist to develop "action plans" to pursue rewarding social activities of their choice.
  Interventions: Behavioral: "Engage & Connect" Psychotherapy
- Symptom Review and Psychoeducation (SRP) (Active Comparator): In this intervention, the therapist will review the participant's symptoms and provide literature-based clinical explanations and clarifications about the symptoms, the course, and the causes of depression. In SRP, the therapist reviews the depressed individual's symptoms, and level of information on depression, identifies misconceptions, and guides selection of educational material which could benefit the patient.
  Interventions: Behavioral: Symptom Review and Psychoeducation (SRP)

INTERVENTIONS:
Behavioral: "Engage & Connect" Psychotherapy — 9-weeks of weekly psychotherapy sessions focused on social reward exposure
  Arms: "Engage & Connect" Psychotherapy
Behavioral: Symptom Review and Psychoeducation (SRP) — 9-weeks of weekly psychotherapy sessions focused on symptom review and psychoeducation about depression and aging
  Arms: Symptom Review and Psychoeducation (SRP)

SUMMARY:
Abnormalities in the Positive Valence System (PVS) are associated with depressive symptoms and reduced behavioral activation in mid- and late-life. This study will investigate the engagement of the PVS during exposure to social rewards, part of a novel streamlined psychotherapy for mid- and late-life depression. Use of computational modeling will enable identification of neuroimaging and behavioral profiles associated with greater treatment response, and may guide future personalization of psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ages aged 50-85 [stratified so that 50% are older than 65]
2. Diagnosis of unipolar major depressive disorder without psychotic features, determined by the SCID
3. Montgomery-Åsberg Depression Rating Scale (MADRS) score ≥ 20.
4. Mini Mental Status Exam (MMSE) ≤ 1 SD below the mean score for patient's age and education
5. Off antidepressants or on a stable dose of an antidepressant for 8 weeks and do not intend to change the dose in the next 10 weeks.
6. Capacity to provide written consent for research assessment and treatment.

Exclusion Criteria:

1. Intent or plan to attempt suicide in the near future.
2. History or presence of psychiatric diagnoses other than major depressive disorder without psychotic features, generalized anxiety disorder, or specific phobia.
3. Use of psychotropic drugs or cholinesterase inhibitors other than use of ≤ 0.5 mg of lorazepam daily up to seven times per week.
4. Neurological disorders (dementias, history of stroke, multiple sclerosis, Parkinson's disease, epilepsy, etc.); cardiac, renal, or respiratory failure; severe chronic obstructive pulmonary disease; metastatic cancer; or debilitated states or less common medical illnesses that may either influence brain systems of interest or ability to participate in the study. Dr. Alexopoulos or another research psychiatrist will review any medical illnesses that does not appear in the list above and determine whether it interferes with the study of positive valence system functions in depression.
5. Contraindications to MRI scanning including cardiac pacemaker, heart valve replacement, vascular stent, insulin pump, cochlear implant, any other metallic biomedical implant contraindicating to MRI, and claustrophobia.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nili Solomonov, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications, after de-identification, as well as study protocol, treatment manuals, statistical analysis plan and informed consent. We will also share our fMRI tasks and analytic code by request with all interested researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After we publish the main results, we will make de-identified data available to other researchers, under a data-sharing agreement overseen by the Weill Cornell ALACRITY Center's Executive Committee.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. All researchers requesting data will commit to using the data solely for research purpose; secure the data; return or destroy it once analyses are completed; do not share it with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | "Engage & Connect" Psychotherapy | Symptom Review and Psychoeducation (SRP)
Started | 31 | 33
Completed | 28 | 30
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Engage & Connect" Psychotherapy | Symptom Review and Psychoeducation (SRP) | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 12 | 15 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 26 | 31 | 57
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 27 | 26 | 53
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting State fMRI Connectivity of the Positive Valence System
Description: Calculated from fMRI scan. Validation of target engagement (resting state functional connectivity (rsFC) within the right hemisphere orbital prefrontal cortex (OFC), specifically between the lateral and medial regions of the OFC).
Time Frame: Baseline, Mid-treatment (Week 5) and Post Treatment (Week 9)
Population: Participants were excluded from analysis in the event no data were collected at baseline due to participant withdrawal, if the participants were clinically excluded during the study, technical issues with MRI data, or lost to follow-up.
Measure: Mean (Standard Error); unit: rsFC correlation coefficient
Arm/Group | "Engage & Connect" Psychotherapy | Symptom Review and Psychoeducation (SRP)
Number analyzed (Participants) | 24 | 23
rsFC correlation coefficient
  Baseline | 0.18 (0.03) | 0.18 (0.02)
  Week 5: number analyzed (Participants) | 23 | 23
  Week 5 | 0.24 (0.02) | 0.29 (0.02)
  Week 9: number analyzed (Participants) | 23 | 23
  Week 9 | 0.25 (0.03) | 0.24 (0.03)
Statistical Analysis 1: Comparison: Symptom Review and Psychoeducation (SRP); Functional connectivity within the orbital prefrontal cortex (OFC; specifically between lateral and medial OFC), significantly changed over time; Test type: Superiority; p = 0.6249, Mixed Models Analysis; Mean Difference (Final Values) = 0.4727

2. Secondary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS)
Description: 10-item Clinician rated measure of depression severity. Scores range from 0 (no depression) to 60 (severe depression).
Time Frame: Baseline, Mid-treatment (Week 5) and Post Treatment (Week 9)
Population: Participants were excluded from analysis in the event no data were collected at baseline due to participant withdrawal, if the participants were clinically excluded during the study, or lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Engage & Connect" Psychotherapy | Symptom Review and Psychoeducation (SRP)
Number analyzed (Participants) | 29 | 31
score on a scale
  Baseline | 23.66 (4.62) | 24.81 (3.39)
  Mid-treatment (Week 5): number analyzed (Participants) | 28 | 29
  Mid-treatment (Week 5) | 13.82 (7.56) | 18.62 (7.03)
  Post Treatment (Week 9): number analyzed (Participants) | 28 | 29
  Post Treatment (Week 9) | 11.86 (8.97) | 14.66 (8.89)
Statistical Analysis 1: Comparison: Symptom Review and Psychoeducation (SRP); Mixed effects model with a fixed effect for treatment and time, as well as time by treatment interaction, and a random effect for subject level. F value for time by treatment interaction; Test type: Superiority; p = .525, Mixed Models Analysis; Mean Difference (Final Values) = 3.8176

3. Secondary Outcome: Change in Behavioral Activation for Depression Scale (BADS)
Description: 25-item measure self-report measure of behavioral activation. Scores range from 0 (very low behavioral activation) to 150 (high behavioral activation).
Time Frame: Baseline, Mid-treatment (Week 5) and Post Treatment (Week 9)
Population: Participants were excluded from analysis in the event no data were collected at baseline due to participant withdrawal, if the participants were clinically excluded during the study, lost to follow-up, or did not complete the BADS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Engage & Connect" Psychotherapy | Symptom Review and Psychoeducation (SRP)
Number analyzed (Participants) | 29 | 31
score on a scale
  Baseline | 71.24 (21.36) | 70.00 (18.40)
  Mid-treatment (Week 5): number analyzed (Participants) | 28 | 29
  Mid-treatment (Week 5) | 95.21 (28.84) | 88.21 (20.73)
  Post Treatment (Week 9): number analyzed (Participants) | 28 | 28
  Post Treatment (Week 9) | 98.00 (30.54) | 93.86 (25.28)
Statistical Analysis 1: Comparison: Symptom Review and Psychoeducation (SRP); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .844, Mixed Models Analysis; Mean Difference (Final Values) = 0.6503

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | "Engage & Connect" Psychotherapy | Symptom Review and Psychoeducation (SRP)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 7/31 | 4/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | "Engage & Connect" Psychotherapy (N=31) | Symptom Review and Psychoeducation (SRP) (N=33)
Wearable device (watch) irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Hospital Visits (unrelated to research) (General disorders) | 4 (4) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04487730/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT04487730/ICF_000.pdf